CLINICAL TRIAL: NCT06048068
Title: Removing Surrogates' Uncertainty to Reduce Fear and Anxiety After Cardiac Events (RESURFACE): A Randomized Pilot Intervention Study
Brief Title: Removing Surrogates' Uncertainty to Reduce Fear and Anxiety After Cardiac Events
Acronym: RESURFACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Sachin Agarwal, Associate Professor of Neurology (Neurocritical Care), Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AAAR8497; P30AG064198 (NIH)
Record Dates: First submitted 2023-09-15; First posted 2023-09-21 (Actual); Results first posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Cardiac Arrest
Keywords: cardiac arrest; uncertainty; cardiac anxiety; acute stress disorder; posttraumatic stress disorder; sleep; caregiver; family; surrogate; information; self care
MeSH Terms: conditions — Heart Arrest; Stress Disorders, Traumatic, Acute; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 2:1 to the informational intervention group or the control group (care as usual). Participants will remain in their assigned arm for the entirety of their study participation. Randomization will be performed using the REDCap randomization module by a study coordinator. This study will be unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Informational Intervention Arm (Experimental): Participants in this arm will receive access to the informational intervention program, via a website link that they will access through their own person phone/tablet/computer.
  Interventions: Behavioral: Educational Informational Platform
- Control Arm (No Intervention): Participants in this arm will receive usual care and no access to the informational intervention program.

INTERVENTIONS:
Behavioral: Educational Informational Platform — This intervention contains many informational articles for surrogates about cardiac arrest, the subsequent hospitalization, and the emotional journey following cardiac arrest. All articles are available in both English and Spanish.
  Other Names: Heartsight website, ourheartsight.com
  Arms: Informational Intervention Arm

SUMMARY:
The goal of this study is to test the feasibility and acceptability of an informational website to reduce uncertainty, psychological distress, and caregiver burden among close family members of cardiac arrest patients. The investigators hypothesize that participants who receive access to the website will have lower rates of uncertainty, psychological distress, and caregiver burden at 3 months post-hospital discharge compared to participants who receive usual care.

DETAILED DESCRIPTION:
This study will be an unblinded, two-arm randomized controlled trial that enrolls up to 100 adult surrogates of living cardiac arrest patients hospitalized in the New York Presbyterian hospital system. Participants must be English- or Spanish-speaking and have a device with internet access. Participants will be randomized 2:1 to receive the informational intervention program or usual care (control).

Intervention arm participants will receive the informational intervention in three discrete packages upon study enrollment, movement to the general medical floor, and at one month post-discharge. All participants will be assessed at study enrollment, hospital discharge, and 3 months post-discharge for their illness uncertainty, psychological distress, and caregiver burden. All participants will also wear a GENEActiv sleep monitor to track their sleep for one week following hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Surrogate of a living NewYork Presbyterian Hospital cardiac arrest patient
* English- or Spanish-speaking
* Has a working smartphone, tablet, laptop, or other device with internet access

Exclusion Criteria:

* Any medical and/or psychiatric impairment precluding them from complying with the protocol
* Non-English and non-Spanish speaking
* Lack of internet/device access
* Surrogate of an adult CA patient who passed away
* Cannot be reached for initial contact (3 unsuccessful attempts made in ICU)
* Moved to the in-patient floor before initial contact can be established

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2023-09-07 (Actual); Primary Completion 2024-10-14 (Actual); Study Completion 2024-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sachin Agarwal, MD, MPH, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center/New York Presbyterian, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sawyer KN, Camp-Rogers TR, Kotini-Shah P, Del Rios M, Gossip MR, Moitra VK, Haywood KL, Dougherty CM, Lubitz SA, Rabinstein AA, Rittenberger JC, Callaway CW, Abella BS, Geocadin RG, Kurz MC; American Heart Association Emergency Cardiovascular Care Committee; Council on Cardiovascular and Stroke Nursing; Council on Genomic and Precision Medicine; Council on Quality of Care and Outcomes Research; and Stroke Council. Sudden Cardiac Arrest Survivorship: A Scientific Statement From the American Heart Association. Circulation. 2020 Mar 24;141(12):e654-e685. doi: 10.1161/CIR.0000000000000747. Epub 2020 Feb 12. PMID 32078390
- [Background] Parnia S, Waller DG, Yeates R, Fenwick P. A qualitative and quantitative study of the incidence, features and aetiology of near death experiences in cardiac arrest survivors. Resuscitation. 2001 Feb;48(2):149-56. doi: 10.1016/s0300-9572(00)00328-2. PMID 11426476
- [Background] van Lommel P, van Wees R, Meyers V, Elfferich I. Near-death experience in survivors of cardiac arrest: a prospective study in the Netherlands. Lancet. 2001 Dec 15;358(9298):2039-45. doi: 10.1016/S0140-6736(01)07100-8. PMID 11755611
- [Background] Azoulay E, Pochard F, Kentish-Barnes N, Chevret S, Aboab J, Adrie C, Annane D, Bleichner G, Bollaert PE, Darmon M, Fassier T, Galliot R, Garrouste-Orgeas M, Goulenok C, Goldgran-Toledano D, Hayon J, Jourdain M, Kaidomar M, Laplace C, Larche J, Liotier J, Papazian L, Poisson C, Reignier J, Saidi F, Schlemmer B; FAMIREA Study Group. Risk of post-traumatic stress symptoms in family members of intensive care unit patients. Am J Respir Crit Care Med. 2005 May 1;171(9):987-94. doi: 10.1164/rccm.200409-1295OC. Epub 2005 Jan 21. PMID 15665319
- [Background] Ann-Britt T, Ella D, Johan H, Asa AB. Spouses' experiences of a cardiac arrest at home: an interview study. Eur J Cardiovasc Nurs. 2010 Sep;9(3):161-7. doi: 10.1016/j.ejcnurse.2009.12.005. Epub 2010 Jan 13. PMID 20071240
- [Background] Grunau B, Dainty K, MacRedmond R, McDonald K, Sasaki A, Sarti AJ, Shemie SD, Cheung A, Gill J. A qualitative exploratory case series of patient and family experiences with ECPR for out-of-hospital cardiac arrest. Resusc Plus. 2021 Apr 28;6:100129. doi: 10.1016/j.resplu.2021.100129. eCollection 2021 Jun. PMID 34223386
- [Background] De Stefano C, Normand D, Jabre P, Azoulay E, Kentish-Barnes N, Lapostolle F, Baubet T, Reuter PG, Javaud N, Borron SW, Vicaut E, Adnet F. Family Presence during Resuscitation: A Qualitative Analysis from a National Multicenter Randomized Clinical Trial. PLoS One. 2016 Jun 2;11(6):e0156100. doi: 10.1371/journal.pone.0156100. eCollection 2016. PMID 27253993
- [Background] Davidson JE, Jones C, Bienvenu OJ. Family response to critical illness: postintensive care syndrome-family. Crit Care Med. 2012 Feb;40(2):618-24. doi: 10.1097/CCM.0b013e318236ebf9. PMID 22080636
- [Background] van Wijnen HG, Rasquin SM, van Heugten CM, Verbunt JA, Moulaert VR. The impact of cardiac arrest on the long-term wellbeing and caregiver burden of family caregivers: a prospective cohort study. Clin Rehabil. 2017 Sep;31(9):1267-1275. doi: 10.1177/0269215516686155. Epub 2017 Jan 9. PMID 28068794
- [Background] Wachelder EM, Moulaert VR, van Heugten C, Verbunt JA, Bekkers SC, Wade DT. Life after survival: long-term daily functioning and quality of life after an out-of-hospital cardiac arrest. Resuscitation. 2009 May;80(5):517-22. doi: 10.1016/j.resuscitation.2009.01.020. Epub 2009 Mar 17. PMID 19282084
- [Background] Douma MJ, Graham TAD, Ali S, Dainty KN, Bone A, Smith KE, Dennet L, Brindley PG, Kroll T, Frazer K. What are the care needs of families experiencing cardiac arrest?: A survivor and family led scoping review. Resuscitation. 2021 Nov;168:119-141. doi: 10.1016/j.resuscitation.2021.09.019. Epub 2021 Sep 27. PMID 34592400
- [Background] Rojas DA, DeForge CE, Abukhadra SL, Farrell L, George M, Agarwal S. Family experiences and health outcomes following a loved ones' hospital discharge or death after cardiac arrest: A scoping review. Resusc Plus. 2023 Mar 3;14:100370. doi: 10.1016/j.resplu.2023.100370. eCollection 2023 Jun. PMID 36909925
- [Background] Bremer A, Dahlberg K, Sandman L. Experiencing out-of-hospital cardiac arrest: significant others' lifeworld perspective. Qual Health Res. 2009 Oct;19(10):1407-20. doi: 10.1177/1049732309348369. PMID 19805803
- [Background] Armand S, Wagner MK, Ozenne B, Verbunt J, Sep SJS, Berg SK, Knudsen GM, Stenbaek DS. Acute Traumatic Stress Screening Can Identify Patients and Their Partners at Risk for Posttraumatic Stress Disorder Symptoms After a Cardiac Arrest: A Multicenter Prospective Cohort Study. J Cardiovasc Nurs. 2021 Aug 16. doi: 10.1097/JCN.0000000000000829. Online ahead of print. PMID 34406981
- [Background] Case R, Stub D, Mazzagatti E, Pryor H, Mion M, Ball J, Cartledge S, Keeble TR, Bray JE, Smith K. The second year of a second chance: Long-term psychosocial outcomes of cardiac arrest survivors and their family. Resuscitation. 2021 Oct;167:274-281. doi: 10.1016/j.resuscitation.2021.06.018. Epub 2021 Jul 6. PMID 34242735
- [Background] Muehlschlegel S, Perman SM, Elmer J, Haggins A, Teixeira Bailey ND, Huang J, Jansky L, Kirchner J, Kasperek-Wynn R, Lipman PD, Yeatts SD, Fetters MD, Dickert NW, Silbergleit R. The Experiences and Needs of Families of Comatose Patients After Cardiac Arrest and Severe Neurotrauma: The Perspectives of National Key Stakeholders During a National Institutes of Health-Funded Workshop. Crit Care Explor. 2022 Mar 4;4(3):e0648. doi: 10.1097/CCE.0000000000000648. eCollection 2022 Mar. PMID 35265851
- [Background] Agarwal S CJ, Newman M, Abukhadra SL, Rojas D, DeForge C, Tincher I, Wylie J, Anderson ML, Marchionda C. . Prioritizing Interventions to Reduce anxiety and posttraumatic stress Among Racially and Ethnically Diverse family surrogates of Cardiac Arrest Survivors in the United States: A Cross-sectional Survey Study. (Under Review). 2022.
- [Background] Anderson EC, Carleton RN, Diefenbach M, Han PKJ. The Relationship Between Uncertainty and Affect. Front Psychol. 2019 Nov 12;10:2504. doi: 10.3389/fpsyg.2019.02504. eCollection 2019. PMID 31781003
- [Background] Bailey DE Jr, Barroso J, Muir AJ, Sloane R, Richmond J, McHutchison J, Patel K, Landerman L, Mishel MH. Patients with chronic hepatitis C undergoing watchful waiting: Exploring trajectories of illness uncertainty and fatigue. Res Nurs Health. 2010 Oct;33(5):465-73. doi: 10.1002/nur.20397. PMID 20730869
- [Background] Hilton BA. Perceptions of uncertainty: its relevance to life-threatening and chronic illness. Crit Care Nurse. 1992 Feb;12(2):70-3. No abstract available. PMID 1544309
- [Background] Dudas K, Olsson LE, Wolf A, Swedberg K, Taft C, Schaufelberger M, Ekman I. Uncertainty in illness among patients with chronic heart failure is less in person-centred care than in usual care. Eur J Cardiovasc Nurs. 2013 Dec;12(6):521-8. doi: 10.1177/1474515112472270. Epub 2013 Jan 9. PMID 23303766
- [Background] Bartley N, Napier CE, Butt Z, Schlub TE, Best MC, Biesecker BB, Ballinger ML, Butow P. Cancer Patient Experience of Uncertainty While Waiting for Genome Sequencing Results. Front Psychol. 2021 Apr 22;12:647502. doi: 10.3389/fpsyg.2021.647502. eCollection 2021. PMID 33967906
- [Background] Ben Salah A, DeAngelis BN, al'Absi M. Uncertainty and psychological distress during COVID-19: What about protective factors? Curr Psychol. 2022 May 28:1-8. doi: 10.1007/s12144-022-03244-2. Online ahead of print. PMID 35669208
- [Background] Agnes Moors PCE, Klaus R. Scherer, and Nico H. Frijda. Appraisal Theories of Emotion: State of the Art and Future Development. Emotion Review 2013 5:2, 119-124. 2013.
- [Background] Chow KM, Chan CW, Chan JC, Choi KK, Siu KY. A feasibility study of a psychoeducational intervention program for gynecological cancer patients. Eur J Oncol Nurs. 2014 Aug;18(4):385-92. doi: 10.1016/j.ejon.2014.03.011. Epub 2014 Apr 30. PMID 24793004
- [Background] Chow KM, H Chan CW, Chan JC. Effects of psychoeducational interventions on sexual functioning, quality of life and psychological outcomes in patients with gynaecological cancer: A systematic review. JBI Libr Syst Rev. 2012;10(58):4077-4164. doi: 10.11124/jbisrir-2012-406. PMID 27820522
- [Background] Nelson EL, Wenzel LB, Osann K, Dogan-Ates A, Chantana N, Reina-Patton A, Laust AK, Nishimoto KP, Chicz-DeMet A, du Pont N, Monk BJ. Stress, immunity, and cervical cancer: biobehavioral outcomes of a randomized clinical trial [corrected]. Clin Cancer Res. 2008 Apr 1;14(7):2111-8. doi: 10.1158/1078-0432.CCR-07-1632. PMID 18381952
- [Background] Levine EG, Silver B. A pilot study: evaluation of a psychosocial program for women with gynecological cancers. J Psychosoc Oncol. 2007;25(3):75-98. doi: 10.1300/J077v25n03_05. PMID 19341015
- [Background] Mishel MH. The measurement of uncertainty in illness. Nurs Res. 1981 Sep-Oct;30(5):258-63. PMID 6912987
- [Background] Eifert GH, Thompson RN, Zvolensky MJ, Edwards K, Frazer NL, Haddad JW, Davig J. The cardiac anxiety questionnaire: development and preliminary validity. Behav Res Ther. 2000 Oct;38(10):1039-53. doi: 10.1016/s0005-7967(99)00132-1. PMID 11004742
- [Background] Weathers F, Litz B, Keane T, Palmieri P, Marx B, Schnurr P. The PTSD checklist for DSM- 5 (PCL-5) Boston. MA: National Center for PTSD. 2013.
- [Background] GENEActiv. Activinsights Ltd. https://www.activinsights.com/products/geneactiv/. Published 2017. Accessed November 21, 2017.
- [Background] Kitko L, McIlvennan CK, Bidwell JT, Dionne-Odom JN, Dunlay SM, Lewis LM, Meadows G, Sattler ELP, Schulz R, Stromberg A; American Heart Association Council on Cardiovascular and Stroke Nursing; Council on Quality of Care and Outcomes Research; Council on Clinical Cardiology; and Council on Lifestyle and Cardiometabolic Health. Family Caregiving for Individuals With Heart Failure: A Scientific Statement From the American Heart Association. Circulation. 2020 Jun 2;141(22):e864-e878. doi: 10.1161/CIR.0000000000000768. Epub 2020 Apr 30. PMID 32349542
- [Background] Johnson CC, Suchyta MR, Darowski ES, Collar EM, Kiehl AL, Van J, Jackson JC, Hopkins RO. Psychological Sequelae in Family Caregivers of Critically III Intensive Care Unit Patients. A Systematic Review. Ann Am Thorac Soc. 2019 Jul;16(7):894-909. doi: 10.1513/AnnalsATS.201808-540SR. PMID 30950647
- [Background] Presciutti A, Newman MM, Grigsby J, Vranceanu AM, Shaffer JA, Perman SM. Associations between posttraumatic stress symptoms and quality of life in cardiac arrest survivors and informal caregivers: A pilot survey study. Resusc Plus. 2021 Feb 4;5:100085. doi: 10.1016/j.resplu.2021.100085. eCollection 2021 Mar. PMID 34223351
- [Background] Van't Wout Hofland J, Moulaert V, van Heugten C, Verbunt J. Long-term quality of life of caregivers of cardiac arrest survivors and the impact of witnessing a cardiac event of a close relative. Resuscitation. 2018 Jul;128:198-203. doi: 10.1016/j.resuscitation.2018.03.016. Epub 2018 Mar 19. PMID 29567463
- [Background] Larsson IM, Wallin E, Rubertsson S, Kristoferzon ML. Relatives' experiences during the next of kin's hospital stay after surviving cardiac arrest and therapeutic hypothermia. Eur J Cardiovasc Nurs. 2013 Aug;12(4):353-9. doi: 10.1177/1474515112459618. Epub 2012 Sep 14. PMID 22984190
- [Background] Wallin E, Larsson IM, Rubertsson S, Kristoferzon ML. Relatives' experiences of everyday life six months after hypothermia treatment of a significant other's cardiac arrest. J Clin Nurs. 2013 Jun;22(11-12):1639-46. doi: 10.1111/jocn.12112. Epub 2013 Feb 28. PMID 23444838
- [Background] Larsen MK, Mikkelsen R, Budin SH, Lamberg DN, Thrysoe L, Borregaard B. With Fearful Eyes: Exploring Relatives' Experiences With Out-of-Hospital Cardiac Arrest: A Qualitative Study. J Cardiovasc Nurs. 2023 Jan-Feb 01;38(1):E12-E19. doi: 10.1097/JCN.0000000000000893. Epub 2022 Jan 7. PMID 35090152
- [Background] Rosenkilde S, Missel M, Wagner MK, Dichman C, Hermansen AS, Larsen MK, Joshi VL, Zwisler AD, Borregaard B. Caught between competing emotions and tensions while adjusting to a new everyday life: a focus group study with family caregivers of out-of-hospital cardiac arrest survivors. Eur J Cardiovasc Nurs. 2023 Apr 12;22(3):320-327. doi: 10.1093/eurjcn/zvac056. PMID 35801906
- [Background] Mion M, Case R, Smith K, Lilja G, Blennow Nordstrom E, Swindell P, Nikolopoulou E, Davis J, Farrell K, Gudde E, Karamasis GV, Davies JR, Toff WD, Abella BS, Keeble TR. Follow-up care after out-of-hospital cardiac arrest: A pilot study of survivors and families' experiences and recommendations. Resusc Plus. 2021 Jul 29;7:100154. doi: 10.1016/j.resplu.2021.100154. eCollection 2021 Sep. PMID 34386781
- [Background] Dougherty CM, Pyper GP, Benoliel JQ. Domains of concern of intimate partners of sudden cardiac arrest survivors after ICD implantation. J Cardiovasc Nurs. 2004 Jan-Feb;19(1):21-31. doi: 10.1097/00005082-200401000-00006. PMID 14994779
- [Background] Pusswald G, Fertl E, Faltl M, Auff E. Neurological rehabilitation of severely disabled cardiac arrest survivors. Part II. Life situation of patients and families after treatment. Resuscitation. 2000 Nov;47(3):241-8. doi: 10.1016/s0300-9572(00)00240-9. PMID 11114453
- [Background] Simons LH, Cunningham S, Catanzaro M. Emotional responses and experiences of wives of men who survive a sudden cardiac death event. Cardiovasc Nurs. 1992 May-Jun;28(3):17-22. No abstract available. PMID 1643654
- [Background] Aggarwal B, Liao M, Christian A, Mosca L. Influence of caregiving on lifestyle and psychosocial risk factors among family members of patients hospitalized with cardiovascular disease. J Gen Intern Med. 2009 Jan;24(1):93-8. doi: 10.1007/s11606-008-0852-1. Epub 2008 Nov 8. PMID 18998190
- [Background] St-Onge MP, Grandner MA, Brown D, Conroy MB, Jean-Louis G, Coons M, Bhatt DL; American Heart Association Obesity, Behavior Change, Diabetes, and Nutrition Committees of the Council on Lifestyle and Cardiometabolic Health; Council on Cardiovascular Disease in the Young; Council on Clinical Cardiology; and Stroke Council. Sleep Duration and Quality: Impact on Lifestyle Behaviors and Cardiometabolic Health: A Scientific Statement From the American Heart Association. Circulation. 2016 Nov 1;134(18):e367-e386. doi: 10.1161/CIR.0000000000000444. Epub 2016 Sep 19. PMID 27647451
- [Background] Moulaert VR, van Heugten CM, Winkens B, Bakx WG, de Krom MC, Gorgels TP, Wade DT, Verbunt JA. Early neurologically-focused follow-up after cardiac arrest improves quality of life at one year: A randomised controlled trial. Int J Cardiol. 2015 Aug 15;193:8-16. doi: 10.1016/j.ijcard.2015.04.229. Epub 2015 Apr 30. PMID 26005166
- [Background] Mishel MH, Braden CJ. Finding meaning: antecedents of uncertainty in illness. Nurs Res. 1988 Mar-Apr;37(2):98-103, 127. PMID 3347527
- [Background] Afifi WA, Felix ED, Afifi TD. The impact of uncertainty and communal coping on mental health following natural disasters. Anxiety Stress Coping. 2012 May;25(3):329-47. doi: 10.1080/10615806.2011.603048. Epub 2011 Aug 1. PMID 21801075
- [Background] Eastwood JA, Doering L, Roper J, Hays RD. Uncertainty and health-related quality of life 1 year after coronary angiography. Am J Crit Care. 2008 May;17(3):232-42; quiz 243. PMID 18450680
- [Background] Penrod J. Refinement of the concept of uncertainty. J Adv Nurs. 2001 Apr;34(2):238-45. doi: 10.1046/j.1365-2648.2001.01750.x. PMID 11430286
- [Background] Sweeny K. On the Experience of Awaiting Uncertain News. Current Directions in Psychological Science. 2018;27(4):281-285.
- [Background] Mishel MH. Uncertainty in chronic illness. Annu Rev Nurs Res. 1999;17:269-94. PMID 10418661
- [Background] Grupe DW, Nitschke JB. Uncertainty and anticipation in anxiety: an integrated neurobiological and psychological perspective. Nat Rev Neurosci. 2013 Jul;14(7):488-501. doi: 10.1038/nrn3524. PMID 23783199
- [Background] Cornelius T, Agarwal S, Garcia O, Chaplin W, Edmondson D, Chang BP. Development and Validation of a Measure to Assess Patients' Threat Perceptions in the Emergency Department. Acad Emerg Med. 2018 Oct;25(10):1098-1106. doi: 10.1111/acem.13513. PMID 29972892
- [Background] Enhancing recovery in coronary heart disease patients (ENRICHD): study design and methods. The ENRICHD investigators. Am Heart J. 2000 Jan;139(1 Pt 1):1-9. doi: 10.1016/s0002-8703(00)90301-6. PMID 10618555
- [Background] National Center for PTSD. PTSD Checklist for DSM-5 (PCL-5). https://www.ptsd.va.gov/professional/assessment/adult-sr/ptsd-checklist.asp. Published February 22, 2018. Accessed2018.
- [Background] Buhr K, Dugas MJ. The Intolerance of Uncertainty Scale: psychometric properties of the English version. Behav Res Ther. 2002 Aug;40(8):931-45. doi: 10.1016/s0005-7967(01)00092-4. PMID 12186356
- [Background] van Hees VT, Sabia S, Anderson KN, Denton SJ, Oliver J, Catt M, Abell JG, Kivimaki M, Trenell MI, Singh-Manoux A. A Novel, Open Access Method to Assess Sleep Duration Using a Wrist-Worn Accelerometer. PLoS One. 2015 Nov 16;10(11):e0142533. doi: 10.1371/journal.pone.0142533. eCollection 2015. PMID 26569414
- [Background] te Lindert BH, Van Someren EJ. Sleep estimates using microelectromechanical systems (MEMS). Sleep. 2013 May 1;36(5):781-9. doi: 10.5665/sleep.2648. PMID 23633761
- [Background] Moore CG, Carter RE, Nietert PJ, Stewart PW. Recommendations for planning pilot studies in clinical and translational research. Clin Transl Sci. 2011 Oct;4(5):332-7. doi: 10.1111/j.1752-8062.2011.00347.x. PMID 22029804
- [Background] Lancaster GA, Dodd S, Williamson PR. Design and analysis of pilot studies: recommendations for good practice. J Eval Clin Pract. 2004 May;10(2):307-12. doi: 10.1111/j..2002.384.doc.x. PMID 15189396

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Informational Intervention Arm | Control Arm
Started | 36 | 17
Completed | 21 | 11
Not Completed | 15 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Informational Intervention Arm | Control Arm | Total
Number analyzed (Participants) | 36 | 17 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 15 | 45
  >=65 years | 6 | 2 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.2 (16.0) | 48.0 (12.6) | 48.2 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 12 | 38
  Male | 10 | 5 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 4 | 12
  Not Hispanic or Latino | 28 | 12 | 40
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 1 | 9
  White | 20 | 10 | 30
  More than one race | 6 | 2 | 8
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 36 | 17 | 53

OUTCOME MEASURES:

1. Primary Outcome: Mishel Uncertainty in Illness Scale Score - Family Member Form
Description: This metric is a 31-item scale measuring surrogates' self-reported uncertainty related to their loved one's cardiac arrest. Participants will be asked to answer from a scale of 1 to 5, 1 being 'Strongly Disagree' and 5 being 'Strongly Agree.' The scale will be scored out of 155. A higher score indicates a greater level of uncertainty.
Time Frame: Data was collected at study enrollment in the ICU (baseline), at hospital discharge (approximately 21 days after baseline), and 3 months post-hospital discharge. The data at 3 months post-discharge is reported
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Informational Intervention Arm | Control Arm
Number analyzed (Participants) | 21 | 11
score on a scale | 82.67 [78.31 to 87.02] | 88.18 [83.04 to 93.32]

2. Secondary Outcome: Post-Traumatic Stress Disorder Checklist (PCL-5) Score
Description: This metric is a 20-item measure of self-reported post-traumatic stress symptoms as defined by the DSM-5. Participants will be asked to score their answer from 0 to 4, 0 being 'Not at all,' and 4 being 'Extremely.' The total score will be out of 80. A higher score indicates more severe PTSD symptoms.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Informational Intervention Arm | Control Arm
Number analyzed (Participants) | 21 | 11
score on a scale | 22.1 (13.3) | 32.7 (12.65)

3. Secondary Outcome: Cardiac Anxiety Questionnaire Score - Fear Subscale
Description: This 8-item metric measures surrogates' self-reported fear of their loved one's cardiac-related stimuli and sensations due to perceived negative consequences. Participants will be asked to rank answers from 1 to 5, 1 being 'Never' and 5 being 'Always.' The total will be out of 40. A higher score indicates more fear and worry related to the heart.
Time Frame: Data was collected at hospital discharge (approximately 21 days after baseline) and 3 months post-hospital discharge. The data at 3 months post-discharge is reported
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Arm | Informational Intervention Arm
Number analyzed (Participants) | 22 | 11
score on a scale | 18.3 (3.8) | 18.9 (7.7)

4. Secondary Outcome: Zarit Burden Interview 12-item Short Form Score
Description: This 12-item metric measures surrogates' self-reported caregiver burden. Participants will be asked to score their answers from 0 to 4, 0 being "Never," and 4 being "Always." The total score is taken out of 48. A higher total score indicates a greater degree of caregiver burden.
Time Frame: At 3 months post-discharge.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Informational Intervention Arm | Control Arm
Number analyzed (Participants) | 22 | 11
score on a scale | 12.5 (6.75) | 18.6 (8.3)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Informational Intervention Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 11/36 | 5/17
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/17
Other Adverse Events (participants affected / at risk) | 0/36 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-10-07): https://cdn.clinicaltrials.gov/large-docs/68/NCT06048068/Prot_SAP_000.pdf